CLINICAL TRIAL: NCT00001622
Title: Study of the Relation Between In Vivo and In Vitro Response of Human Small Vessels
Brief Title: Study of the Response of Human Small Blood Vessels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970098; 97-H-0098
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Healthy; Hypercholesterolemia; Hypertension
Keywords: Endothelium; Hypercholesterolemia; Hypertension; Microvessels; Vasodilation; Normal Volunteer
MeSH Terms: conditions — Hypercholesterolemia; Hypertension; Aneurysm

INTERVENTIONS:
Procedure: investigate the relationship between in vivo and in vitro vascular responses

SUMMARY:
A layer of cells called the endothelium line the walls of blood vessels. These cells produce substances that control the tone of blood vessels and thus control blood flow through the vessel. One of the substances produced involved in the control of blood vessel function is nitric oxide. Nitric oxide (NO) plays a role in the relaxation of blood vessels.

Researchers have been interested in the function of the endothelium in patients with high blood pressure (essential hypertension) and patients with high cholesterol (hypercholesterolemia).

After conducting studies on the endothelium and nitric oxide, researchers have found that the endothelium is indeed functioning abnormally in patients with high blood pressure and high cholesterol. In addition, researchers have determined that the dysfunction is a result of abnormalities in the nitric oxide (NO) system.

In this study researchers plan to investigate the relationship between blood vessel responses in real-life settings versus laboratory settings in normal volunteers, patients with high blood pressure, and patients with high cholesterol.

DETAILED DESCRIPTION:
Over the last ten years, we have been interested in the investigation of endothelial function in patients with essential hypertension and patients with hypercholesterolemia. We have performed intra-arterial infusion of endothelium-dependent and endothelium-independent drugs into the brachial artery with noninvasive measurement of the response of the forearm vasculature by means of strain gauge plethysmography. Those studies have allowed us to: a) demonstrate the presence of endothelial dysfunction in patients with essential hypertension and in patients with hypercholesterolemia; and b) identify an abnormality in the endothelium-derived nitric oxide system that is responsible for endothelial dysfunction in these patients. Further studies to more precisely determine the intracellular processes that mediate this abnormality in endothelial function in these patients are limited by the inherent shortcomings of the in vivo technique. An alternative possibility is the study of human small vessels in vitro; however, the relationship between in vivo and in vitro vascular responses to endothelium-dependent and -independent agonists has not been established. In the present study, we propose to investigate this relationship in normal volunteers, patients with essential hypertension, and patients with hypercholesterolemia.

ELIGIBILITY:
Patients (men and nonpregnant women) with systemic hypertension, patients with hypercholesterolemia, and normal volunteers.

All blood pressure recordings must be consistently elevated.

No renovascular hypertension or other etiologies for elevated blood pressure.

No definite evidence of accelerated or malignant hypertension (diastolic pressures above 115 mmHg, with associated encephalopathic changes, papilledema, progressive renal failure, or congestive heart failure), or serious intercurrent illness.

Patients in whom withdrawal of antihypertensive medications is considered hazardous are ineligible.

Patients in whom the blood pressure remains at normal levels 2 weeks after withdrawal of antihypertensive treatment will be closely monitored until they become hypertensive, at which time they will undergo the study. Patients in whom blood pressure does not increase after 2 months of discontinuation of therapy will be excluded from the study.

Patients with coexistent hypertension and hypercholesterolemia are ineligible.

Normal volunteers who are not taking any kind of medication are eligible.

No history of diabetes, peripheral vascular disease, coagulopathy, or any other disease predisposing to vasculitis or Raynaud's phenomenon.

No history of keloid formation.

All patients must be capable of giving informed consent for all procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 87
Dates: Start 1997-03; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Furchgott RF. Role of endothelium in responses of vascular smooth muscle. Circ Res. 1983 Nov;53(5):557-73. doi: 10.1161/01.res.53.5.557. No abstract available. PMID 6313250
- [Background] Falloon BJ, Heagerty AM. In vitro perfusion studies of human resistance artery function in essential hypertension. Hypertension. 1994 Jul;24(1):16-23. doi: 10.1161/01.hyp.24.1.16. PMID 8021003
- [Background] Goode GK, Heagerty AM. In vitro responses of human peripheral small arteries in hypercholesterolemia and effects of therapy. Circulation. 1995 Jun 15;91(12):2898-903. doi: 10.1161/01.cir.91.12.2898. PMID 7796498